CLINICAL TRIAL: NCT02908308
Title: Targeted Hypothermia Versus Targeted Normothermia After Out-of-hospital Cardiac Arrest (TTM2) - A Randomised Clinical Trial
Brief Title: Targeted Hypothermia Versus Targeted Normothermia After Out-of-hospital Cardiac Arrest
Acronym: TTM-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helsingborgs Hospital (Other)
Collaborators: Lund University (Other); Region Skåne - Skånevård SUND (Unknown); Copenhagen Trial Unit, Center for Clinical Intervention Research (Other); Clinical Trials Sweden, Forum South (Unknown); Integrated Biobank of Luxembourg (Other)
Responsible Party: Principal Investigator, Niklas Nielsen, MD, PhD, Associate professor, Helsingborgs Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TTM-2
Record Dates: First submitted 2016-09-16; First posted 2016-09-20 (Estimated); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Out-of-hospital Cardiac Arrest
Keywords: Induced hypothermia; Mild induced hypothermia; Therapeutic hypothermia; Cardiac arrest; Out-of-hospital cardiac arrest; Mortality; Neurological function; Randomised clinical trial
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Heart Arrest | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The clinical team responsible for the participant (physicians, nurses and others) and involved with direct patient care will not be blinded to allocation group due to the inherent difficulty in blinding the intervention and as temperature is a vital sign required for clinical care. Measures will be taken to ensure that the information about allocation will not disseminate beyond the immediate group of caregivers responsible for patient care. A blinded physician will evaluate the patient at 96 hours after randomisation and make a statement on neurological prognosis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normothermia (Active Comparator): Standard care with early treatment of fever. Active temperature control with a device will be used if the patient develops a temperature greater than or equal 37.8°C.
  Interventions: Procedure: Standard care with early treatment of fever
- Hypothermia (Experimental): Targeted temperature management to 33°C for up to 28h.
  Interventions: Procedure: Targeted temperature management to 33°C

INTERVENTIONS:
Procedure: Targeted temperature management to 33°C — Rapid cooling to below 33°C, followed by temperature control at 33°C for up to 28h.
  Arms: Hypothermia
Procedure: Standard care with early treatment of fever — Normothermia and standard care - use of a device for temperature control if temperature is greater than or equal to 37.8°C
  Arms: Normothermia

SUMMARY:
ILCOR guidelines recommend Target Temperature Management (TTM) to between 32°C and 36°C after out-of-hospital cardiac arrest, based on low quality evidence. In a previous trial, TTM at 33°C did not confer a survival benefit or improved neurological function, compared to TTM at 36°C. A lower target temperature might be beneficial compared with normothermia and early treatment of fever. Therefore the primary purpose of the TTM2-trial will be to study any differences in mortality, neurological function and quality of life between a target temperature of 33°C and standard care avoiding fever.

DETAILED DESCRIPTION:
The TTM2 trial is a continuation of the collaboration that resulted in the previous Targeted Temperature Management after out-of-hospital cardiac arrest trial (hereafter: TTM1). With its planned size with it will supersede the TTM1 trial as the largest trial on temperature management as a post-cardiac arrest treatment.

The TTM1 trial (NCT01020916) was a multicenter, multinational, outcome assessor-blinded, parallel group, randomised clinical trial comparing two strict target temperature regimens of 33°C and 36°C in adult patients, who have sustained return of spontaneous circulation and are unconscious after out-of-hospital cardiac arrest, when admitted to hospital. The trial did not demonstrate any difference in survival until end of trial (Hazard Ratio with a point estimate in favour of 36°C of 1.06 (95% confidence interval 0.89-1.28; P=0.51) or neurologic function at six months after the arrest, measured with CPC and mRS.

The planned study is a international, multicenter, parallel group, non-commerical, randomized, superiority trial in which a target temperature om 33°C after cardiac arrest will be compared to normothermia and early treatment of fever.

Patients eligible for inclusion will be unconscious adult patients with OHCA of a presumed cardiac cause with stable return of spontaneous circulation. Randomization will be performed by a physician in the emergency department, in the angiography suite or in the intensive care unit via web-based application using permuted blocks with varying sizes, stratified by site. Due to the nature of the intervention, health care staff will not be blinded to the intervention. However, the physicians who will assess outcomes will be blinded to temperature allocation, as will those who perform prognostication.

The intervention period will commence at the time of randomization. Cooling in the hypothermia group will achieved by means of cold fluids and state-of-the-art cooling devices (intravascular or body-surface applied closed loop systems). The initial aim will be to achieve a body temperature of 33.0°C. When this has been achieved, the target temperature will be 33°C until 28 hours after randomisation. When 28 hours have passed, gradual rewarming at a rate of 1/3°C per hour will commence, this will allow 12 hours for rewarming.

In the normothermia arm the aim will be to avoid a temperature greater than or equal to 37.8°C using conservative measures. If a single temperature of 37.8° or greater is measured, active cooling with a device should be initiated and maintained until 40 hours after randomization.

All participants will be sedated, mechanically ventilated and hemodynamically supported throughout the intervention period of 40 hours. Participants in both arms who remain comatose after 40h should be kept at a normothermic level (36.5 - 37.7°C) until 72h after randomization and active warming should be avoided.

Participants who remain unconscious four days after randomization will be assessed according to a conservative protocol based on the European Resuscitation Council's recommendations for withdrawal of life sustaining therapies.

Follow up will be performed at:

1 month (face-to-face or telephone), Assessment according to the modified Rankin scale (mRS)

6 moths (face-to-face), Assessment according to the mRS-scale. Assessment of health-related quality of life using EQ5D-5L.

ELIGIBILITY:
Inclusion Criteria:

* Out-of-hospital cardiac arrest
* Presumed cardiac cause of cardiac arrest
* Unconscious with a FOUR-score <M4 (not obeying verbal commands)
* Stable return of spontaneous circulation (20 min)
* Eligible for intensive care treatment without restrictions
* Inclusion within 180 minutes of ROSC

Exclusion Criteria:

* Unwitnessed cardiac arrest with an initial rhythm of asystole
* Temperature on admission <30°C.
* On ECMO prior to ROSC
* Obvious or suspected pregnancy
* Intracranial bleeding
* On ECMO prior to ROSC
* Severe chronic obstructive pulmonary disorder (COPD) with long-term home oxygen therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1900 (Actual)
Dates: Start 2017-11-18 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Mortality | 180 days
  Landmark mortality at 180 days

SECONDARY OUTCOMES:
Poor functional outcome | 180 days
  Assessed using the modified Rankin Scale (mRS), with a score of 4-6 being a poor outcome.
Days alive outside hospital | 180 days.
  Number of days alive within 180 days from initial hospital discharge.
Quality of Life | 180 days
  Health-related Quality of Life - EQ-5D (VAS scale)
Quality of Life | 180 days
  Health-related Quality of Life - EQ-5D (Index value)
Survival until end of the trial | 180 days after randmomization of the last patient
  Mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Niklas Nielsen, MD, PhD, Principal Investigator — Helsingborgs lasarett, Region Skåne, Sweden; Hans Friberg, MD, PhD, Principal Investigator — Lund University Hospital, Lund, Sweden; Tobias Cronberg, MD, PhD, Principal Investigator — Lund University Hospital, Lund, Sweden; Jan Hovdenes, MD, PhD, Principal Investigator — Oslo University Hospital, Oslo, Norway; Matt P Wise, MD, PhD, Principal Investigator — University Hospital of Wales, Cardiff, UK; Clifton W Callaway, MD, PhD, Principal Investigator — University of Pittsburgh, Pittsburgh, USA; Christian Storm, MD, PhD, Principal Investigator — Charité-University Medicine (Berlin, Germany); Alain Cariou, MD, PhD, Principal Investigator — Université Paris Descartes, France; David Erlinge, MD, PhD, Principal Investigator — Lund University Hospital, Lund, Sweden; Christian Rylander, MD, PhD, Principal Investigator — Sahlgrenska University Hospital; Josef Dankiewicz, MD, PhD, Principal Investigator — Skåne University Hospital Lund; Mauro Oddo, MD, PhD, Principal Investigator — Université de Lausanne, Lausanne, Switzerland; Manoj Saxena, MD, PhD, Principal Investigator — The George Institute for Global Health (Sydney, Australia); Per Nordberg, MD, PhD, Principal Investigator — Södersjukhuset, Stockholm; Fabio Taccone, MD, PhD, Principal Investigator — Hopital Erasme, Brussles, Belgium; Paolo Pelosi, MD, PhD, Principal Investigator — San Martino University Hospital, Genoa; Michael Ioannidis, MD, PhD, Principal Investigator — Innsbruck University Hospital; Jan Belholavek, MD, PhD, Principal Investigator — Prague University Hospital; Paul Young, MD, Principal Investigator — Wellington Regional Hospital; Hans Kirkegaard, MD,PhD, Principal Investigator — Aarhus University Hospital; Alistair Nichol, MD, PhD, Principal Investigator — Department of Anaesthesia and Intensive Care Medicine, St Vincent's University Hospital
Locations (60):
- United States (2):
  - Mayo Clinic Hospital-St. Mary's Campus, Rochester, New York
  - UPMC-Presbyterian, Pittsburgh, Pennsylvania
- Australia (10):
  - John Hunter Hospital, Newcastle, New South Wales
  - Concord Repatriation General Hospital, Sydney, New South Wales
  - Liverpool Hospital, Sydney, New South Wales
  - St Vincent's Hospital, Sydney, New South Wales
  - Princess Alexandra Hospital, Brisbane, Queensland
  - Northern Hospital, Epping, Victoria
  - The Alfred, Melbourne, Victoria
  - Austin Hospital, Melbourne
  - Nepean Hospital, Sydney
  - Royal North Shore Hospital, Sydney
- Innsbruck University Hospital, Innsbruck, Austria
- Belgium (2):
  - Erasme Hospital, Brussels
  - Ziekenhuis Oost-Limburg, Genk
- Czechia (3):
  - Hradec Kralove Hospital, Hradec Králové
  - Liberec Hospital, Liberec
  - General University Hospital, Prague
- Aarhus University Hospital, Aarhus, Denmark
- France (5):
  - Chu Dupuytren, Limoges
  - CHU Nantes, Nantes
  - Cochin University Hospital, Paris
  - Lariboisière Hospital, Paris
  - Versailles Hospital, Versailles
- Charité, Campus Virchow, Berlin, Germany
- Italy (2):
  - San Martino Hospital, Genova
  - Modena NOCSAE Hospital, Modena
- New Zealand (2):
  - Christchurch Hospital, Christchurch
  - Wellington Hospital, Wellington
- Norway (4):
  - Sorlandet Hospital, Arendal
  - Haukeland Hospital, Bergen
  - Oslo University Hospital, Oslo
  - St. Olav's University Hospital, Trondheim
- Sweden (13):
  - Hallands Hospital, Halmstad, Halland County
  - Skane University Hospital - Lund, Lund, Skåne County
  - Skane University Hospital - Malmö, Malmo, Skåne County
  - Sahlgrenska University Hospital, Gothenburg
  - Helsingborgs Hospital, Helsingborg
  - Centralsjukhuset i Karlstad, Karlstad
  - Linköping University Hospital, Linköping
  - Örebro University Hospital, Örebro
  - Skaraborgs sjukhus, Skövde
  - Capio St:Göran, Stockholm
  - Södersjukhuset, Stockholm
  - Norra Älvsborgs Länssjukhus (NÄL), Trollhättan
  - Akademiska Sjukhuset, Uppsala
- Switzerland (5):
  - University Hospital Bern, Inselspital, Bern
  - University Hospital of Lausanne, Lausanne
  - Cardiocentro Ticino, Lugano
  - Kantonsspital St.Gallen, Sankt Gallen
  - Zurich University Hospital, Zurich
- United Kingdom (9):
  - Basildon and Thurrock Hospitals NHS Foundation Trust - Essex CTC, Basildon
  - Royal Victoria Hospital, Belfast
  - Birmingham University Hospital, Birmingham
  - Royal Bournemouth and Christchurch Hospitals NHS Foundation Trust, Bournemouth
  - Bristol Royal Infirmary, Bristol
  - University Hospital of Wales, Cardiff
  - Manchester Royal Infirmary, Manchester
  - Queen Alexandra Hospital, Portsmouth
  - Royal Berkshire Hospital, Reading

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Nielsen N, Wetterslev J, Cronberg T, Erlinge D, Gasche Y, Hassager C, Horn J, Hovdenes J, Kjaergaard J, Kuiper M, Pellis T, Stammet P, Wanscher M, Wise MP, Aneman A, Al-Subaie N, Boesgaard S, Bro-Jeppesen J, Brunetti I, Bugge JF, Hingston CD, Juffermans NP, Koopmans M, Kober L, Langorgen J, Lilja G, Moller JE, Rundgren M, Rylander C, Smid O, Werer C, Winkel P, Friberg H; TTM Trial Investigators. Targeted temperature management at 33 degrees C versus 36 degrees C after cardiac arrest. N Engl J Med. 2013 Dec 5;369(23):2197-206. doi: 10.1056/NEJMoa1310519. Epub 2013 Nov 17. PMID 24237006
- [Derived] Gobel Andertun S, Wissendorff-Ekdahl A, Ullen S, Cronberg T, Friberg H, Jakobsen JC, Blennow Nordstrom E, Heimburg K, Cariou A, Grejs AM, Haenggi M, Hovdenes J, Robba C, Rylander C, Taccone FS, Wise MP, Young PJ, Nielsen N, Lilja G. Impact of frailty on mortality, functional outcome, and health status after out-of-hospital cardiac arrest: insights from the TTM2-trial. Intensive Care Med. 2025 Dec;51(12):2367-2377. doi: 10.1007/s00134-025-08185-5. Epub 2025 Nov 10. PMID 41212202
- [Derived] Admiraal MM, Backman S, Annborn M, Borgquist O, Dankiewicz J, During J, Legriel S, Lilja G, Lindehammer H, Nielsen N, Rossetti AO, Unden J, Cronberg T, Westhall E; TTM2-trial investigators. Electrographic and Clinical Determinants of Good Outcome After Postanoxic Status Epilepticus. Neurology. 2025 Mar 11;104(5):e210304. doi: 10.1212/WNL.0000000000210304. Epub 2025 Feb 11. PMID 39933130
- [Derived] Taccone FS, Cariou A, Zorzi S, Friberg H, Jakobsen JC, Nordberg P, Robba C, Belohlavek J, Hovdenes J, Haenggi M, Aneman A, Grejs A, Keeble TR, Annoni F, Young PJ, Wise MP, Cronberg T, Lilja G, Nielsen N, Dankiewicz J. Hypothermia versus normothermia in patients with cardiac arrest and shockable rhythm: a secondary analysis of the TTM-2 study. Crit Care. 2024 Oct 15;28(1):335. doi: 10.1186/s13054-024-05119-3. PMID 39407230
- [Derived] Heimburg K, Blennow Nordstrom E, Dankiewicz J, Friberg H, Grejs AM, Hanggi M, Keeble TR, Kirkegaard H, Nielsen N, Rylander C, Tornberg AB, Ullen S, Wise MP, Cronberg T, Lilja G. Low physical activity level in out-of-hospital cardiac arrest survivors with obesity, mobility problems and cognitive impairment: Results from the TTM2 trial. Resuscitation. 2024 Nov;204:110407. doi: 10.1016/j.resuscitation.2024.110407. Epub 2024 Oct 4. PMID 39368797
- [Derived] Battaglini D, Schiavetti I, Ball L, Jakobsen JC, Lilja G, Friberg H, Wendel-Garcia PD, Young PJ, Eastwood G, Chew MS, Unden J, Thomas M, Joannidis M, Nichol A, Lundin A, Hollenberg J, Hammond N, Saxena M, Martin A, Solar M, Taccone FS, Dankiewicz J, Nielsen N, Morten Grejs A, Wise MP, Hangghi M, Smid O, Patroniti N, Robba C; TTM2 trial investigators. Association between early airway intervention in the pre-hospital setting and outcomes in out of hospital cardiac arrest patients: A post-hoc analysis of the Target Temperature Management-2 (TTM2) trial. Resuscitation. 2024 Oct;203:110390. doi: 10.1016/j.resuscitation.2024.110390. Epub 2024 Sep 5. PMID 39244144
- [Derived] Lang M, Kenda M, Scheel M, Martola J, Wheeler M, Owen S, Johnsson M, Annborn M, Dankiewicz J, Deye N, During J, Friberg H, Halliday T, Jakobsen JC, Lascarrou JB, Levin H, Lilja G, Lybeck A, McGuigan P, Rylander C, Sem V, Thomas M, Ullen S, Unden J, Wise MP, Cronberg T, Wasselius J, Nielsen N, Leithner C, Moseby-Knappe M. Standardised and automated assessment of head computed tomography reliably predicts poor functional outcome after cardiac arrest: a prospective multicentre study. Intensive Care Med. 2024 Jul;50(7):1096-1107. doi: 10.1007/s00134-024-07497-2. Epub 2024 Jun 20. PMID 38900283
- [Derived] Holgersson J, Meyer MAS, Dankiewicz J, Lilja G, Ullen S, Hassager C, Cronberg T, Wise MP, Belohlavek J, Hovdenes J, Pelosi P, Erlinge D, Schrag C, Smid O, Brunetti I, Rylander C, Young PJ, Saxena M, Aneman A, Cariou A, Callaway C, Eastwood GM, Haenggi M, Joannidis M, Keeble TR, Kirkegaard H, Leithner C, Levin H, Nichol AD, Morgan MPG, Nordberg P, Oddo M, Storm C, Taccone FS, Thomas M, Bro-Jeppesen J, Horn J, Kjaergaard J, Kuiper M, Pellis T, Stammet P, Wanscher MJ, Friberg H, Nielsen N, Jakobsen JC. Hypothermic versus Normothermic Temperature Control after Cardiac Arrest. NEJM Evid. 2022 Nov;1(11):EVIDoa2200137. doi: 10.1056/EVIDoa2200137. Epub 2022 Jun 15. PMID 38319850
- [Derived] Lilja G, Ullen S, Dankiewicz J, Friberg H, Levin H, Nordstrom EB, Heimburg K, Jakobsen JC, Ahlqvist M, Bass F, Belohlavek J, Olsen RB, Cariou A, Eastwood G, Fanebust HR, Grejs AM, Grimmer L, Hammond NE, Hovdenes J, Hrecko J, Iten M, Johansen H, Keeble TR, Kirkegaard H, Lascarrou JB, Leithner C, Lesona ME, Levis A, Mion M, Moseby-Knappe M, Navarra L, Nordberg P, Pelosi P, Quayle R, Rylander C, Sandberg H, Saxena M, Schrag C, Siranec M, Tiziano C, Vignon P, Wendel-Garcia PD, Wise MP, Wright K, Nielsen N, Cronberg T. Effects of Hypothermia vs Normothermia on Societal Participation and Cognitive Function at 6 Months in Survivors After Out-of-Hospital Cardiac Arrest: A Predefined Analysis of the TTM2 Randomized Clinical Trial. JAMA Neurol. 2023 Oct 1;80(10):1070-1079. doi: 10.1001/jamaneurol.2023.2536. PMID 37548968
- [Derived] Robba C, Badenes R, Battaglini D, Ball L, Sanfilippo F, Brunetti I, Jakobsen JC, Lilja G, Friberg H, Wendel-Garcia PD, Young PJ, Eastwood G, Chew MS, Unden J, Thomas M, Joannidis M, Nichol A, Lundin A, Hollenberg J, Hammond N, Saxena M, Martin A, Solar M, Taccone FS, Dankiewicz J, Nielsen N, Grejs AM, Ebner F, Pelosi P; TTM2 Trial collaborators. Oxygen targets and 6-month outcome after out of hospital cardiac arrest: a pre-planned sub-analysis of the targeted hypothermia versus targeted normothermia after Out-of-Hospital Cardiac Arrest (TTM2) trial. Crit Care. 2022 Oct 21;26(1):323. doi: 10.1186/s13054-022-04186-8. PMID 36271410
- [Derived] Lang M, Leithner C, Scheel M, Kenda M, Cronberg T, During J, Rylander C, Annborn M, Dankiewicz J, Deye N, Halliday T, Lascarrou JB, Matthew T, McGuigan P, Morgan M, Thomas M, Ullen S, Unden J, Nielsen N, Moseby-Knappe M. Prognostic accuracy of head computed tomography for prediction of functional outcome after out-of-hospital cardiac arrest: Rationale and design of the prospective TTM2-CT-substudy. Resusc Plus. 2022 Oct 12;12:100316. doi: 10.1016/j.resplu.2022.100316. eCollection 2022 Dec. PMID 36267356
- [Derived] During J, Annborn M, Cariou A, Chew MS, Dankiewicz J, Friberg H, Haenggi M, Haxhija Z, Jakobsen JC, Langeland H, Taccone FS, Thomas M, Ullen S, Wise MP, Nielsen N. Influence of temperature management at 33 degrees C versus normothermia on survival in patients with vasopressor support after out-of-hospital cardiac arrest: a post hoc analysis of the TTM-2 trial. Crit Care. 2022 Jul 31;26(1):231. doi: 10.1186/s13054-022-04107-9. PMID 35909163
- [Derived] Robba C, Badenes R, Battaglini D, Ball L, Brunetti I, Jakobsen JC, Lilja G, Friberg H, Wendel-Garcia PD, Young PJ, Eastwood G, Chew MS, Unden J, Thomas M, Joannidis M, Nichol A, Lundin A, Hollenberg J, Hammond N, Saxena M, Annborn M, Solar M, Taccone FS, Dankiewicz J, Nielsen N, Pelosi P; TTM2 Trial Collaborators. Ventilatory settings in the initial 72 h and their association with outcome in out-of-hospital cardiac arrest patients: a preplanned secondary analysis of the targeted hypothermia versus targeted normothermia after out-of-hospital cardiac arrest (TTM2) trial. Intensive Care Med. 2022 Aug;48(8):1024-1038. doi: 10.1007/s00134-022-06756-4. Epub 2022 Jul 2. PMID 35780195
- [Derived] Robba C, Nielsen N, Dankiewicz J, Badenes R, Battaglini D, Ball L, Brunetti I, Pedro David WG, Young P, Eastwood G, Chew MS, Jakobsen J, Unden J, Thomas M, Joannidis M, Nichol A, Lundin A, Hollenberg J, Lilja G, Hammond NE, Saxena M, Martin A, Solar M, Taccone FS, Friberg HA, Pelosi P. Ventilation management and outcomes in out-of-hospital cardiac arrest: a protocol for a preplanned secondary analysis of the TTM2 trial. BMJ Open. 2022 Mar 3;12(3):e058001. doi: 10.1136/bmjopen-2021-058001. PMID 35241476
- [Derived] Dankiewicz J, Cronberg T, Lilja G, Jakobsen JC, Levin H, Ullen S, Rylander C, Wise MP, Oddo M, Cariou A, Belohlavek J, Hovdenes J, Saxena M, Kirkegaard H, Young PJ, Pelosi P, Storm C, Taccone FS, Joannidis M, Callaway C, Eastwood GM, Morgan MPG, Nordberg P, Erlinge D, Nichol AD, Chew MS, Hollenberg J, Thomas M, Bewley J, Sweet K, Grejs AM, Christensen S, Haenggi M, Levis A, Lundin A, During J, Schmidbauer S, Keeble TR, Karamasis GV, Schrag C, Faessler E, Smid O, Otahal M, Maggiorini M, Wendel Garcia PD, Jaubert P, Cole JM, Solar M, Borgquist O, Leithner C, Abed-Maillard S, Navarra L, Annborn M, Unden J, Brunetti I, Awad A, McGuigan P, Bjorkholt Olsen R, Cassina T, Vignon P, Langeland H, Lange T, Friberg H, Nielsen N; TTM2 Trial Investigators. Hypothermia versus Normothermia after Out-of-Hospital Cardiac Arrest. N Engl J Med. 2021 Jun 17;384(24):2283-2294. doi: 10.1056/NEJMoa2100591. PMID 34133859
- [Derived] Dankiewicz J, Cronberg T, Lilja G, Jakobsen JC, Belohlavek J, Callaway C, Cariou A, Eastwood G, Erlinge D, Hovdenes J, Joannidis M, Kirkegaard H, Kuiper M, Levin H, Morgan MPG, Nichol AD, Nordberg P, Oddo M, Pelosi P, Rylander C, Saxena M, Storm C, Taccone F, Ullen S, Wise MP, Young P, Friberg H, Nielsen N. Targeted hypothermia versus targeted Normothermia after out-of-hospital cardiac arrest (TTM2): A randomized clinical trial-Rationale and design. Am Heart J. 2019 Nov;217:23-31. doi: 10.1016/j.ahj.2019.06.012. Epub 2019 Jun 26. PMID 31473324
- See also: Trial official webpage — http://ttm2trial.org